CLINICAL TRIAL: NCT05323682
Title: Physical Excercise Program in Children With Drug-resistant Epilepsy
Acronym: PEPDRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIB SIM
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy in Children

STUDY DESIGN:
Intervention Model Description: Prospective, experimental, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Individualized physical exercise program
  Interventions: Other: Individualized physical exercise program
- Control (Active Comparator): No individualized physical exercise program
  Interventions: Other: NO Individualized physical exercise program

INTERVENTIONS:
Other: Individualized physical exercise program — An individualized physical exercise program was programmed, monitored remotely by e-mail or the use of an activity wristband
  Arms: Experimental
Other: NO Individualized physical exercise program — Usual medication
  Arms: Control

SUMMARY:
Pediatric epilepsy has been described as an age related-condition, and it has a strong impact on childhood quality of life. Psychological symptoms and self-esteem impairment are common facts. Although there are some studies studying the benefits of physical exercise in order to improve seizure control in adults with epilepsy, we have not found studies that support it in pediatric population. Few studieshave reported in childhood some benefits in terms of quality of life, self-esteem and improvement of neuropsychological symptoms. Therefore, it is necessary to use a validated and applicable scale of quality of life in children with epilepsy. Otherwise, findings may be difficult to reproduce

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-14 years
2. Diagnosis of epilepsy (must meet at least one of the following criteria):

   1. At least 2 unprovoked seizures in a period of more than 24 hours
   2. A seizure and probability of future seizures similar to the general risk of recurrence (60% or more) than if the patient had had 2 crises.
   3. Diagnosis of epileptic syndrome.
3. Adequate communication skills with your family.
4. Absence of significant motor limitation.
5. Parents or legal guardians must have given consent to participate in the study.

Exclusion Criteria:

b) Exclusion criteria:

1. Failure to meet any of the aforementioned requirements.
2. Failure to complete completely and/or legibly any of the instruments of evaluation. c) Abandonment criteria

1. Failure to deliver the submitted questionnaires in a timely manner. 2. Failure to attend the scheduled appointment to complete the questionnaires control. 3. Not responding to phone calls, e-mails or requests made to make a new appointment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
PedsQL (Pediatric Quality of Life Inventory) | Up to 6 months
  Likert scale 0-5
(Quality of Life in Childhood Epilepsy Questionary, QoLCE) | Up to 6 months
  16 items version
PAQ-C (Physical Activity Questionnaire) | Up to 6 months
  Likert scale 0-5
BMI (Body mass index) | Up to 6 months
  (kg)/height (m2)
Waist/hip ratio | Up to 6 months
  ICC= w/h (cm)
Tricipital skinfold | Up to 6 months
  Thickness of the skinfold located over the triceps muscle
Subscapular skinfold | Up to 6 months
  Thickness of localized adipose tissue immediately below the inferior angle of the scapula
Lower extremity strength | Up to 6 months
  Standing Long Jump Test
Grip strength | Up to 6 months
  Takei Tkk 5401 Digital Hand Dynamometer below the inferior angle of the scapula
Cardiorespiratory fitness. | Up to 6 months
  It was carried out with the Course Navette test (round trip 20 meters)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No